CLINICAL TRIAL: NCT04911101
Title: Performance Indicators and Patient Experience in 7G and 10G Vacuum-assisted Excision of Probably Benign Breast Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Stockholm South General Hospital (Other); Capio Sankt Görans Hospital (Other); Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Fredrik Strand, Consultant (biträdande överläkare), Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K2019-7986
Record Dates: First submitted 2021-05-20; First posted 2021-06-02 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Breast Diseases
Keywords: Vacuum-assisted excision; Breast; Minimally invasive procedure; Needle size
MeSH Terms: conditions — Breast Diseases | interventions — Needles

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 7G needle (Experimental): 7G needle dimension used
  Interventions: Device: Excision with 7G needle
- 10G needle (Experimental): 10G needle dimension used
  Interventions: Device: Excision with 10G needle

INTERVENTIONS:
Device: Excision with 7G needle — Vacuum-assisted excision using a biopsy needle with two alternative dimensions
  Arms: 7G needle
Device: Excision with 10G needle — Vacuum-assisted excision using a biopsy needle with two alternative dimensions
  Arms: 10G needle

SUMMARY:
The purpose of this study is to assess how the needle size 7G vs 10G affects performance indicators and patient experience in vacuum-assisted excision (VAE) of probably benign breast lesions

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will have a VAE procedure to remove their breast lesion and will be randomised to either 7G or 10G needle size. After completion of the procedure, the patients fill out a questionnaire to collect data on their experience. The radiologist performing the procedure fills out a form collecting procedural performance indicators.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-verified probably benign breast lesion less than 20 mm size
* Biopsy-verified benign breast lesion less than 30 mm size
* Screen-detected group of microcalcifications under 10 mm size

Exclusion Criteria:

* Age less than 18 years of age
* Inability to understand the meaning of informed consent
* Pregnancy
* Breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Excision time | Baseline
  Time from excision start to excision stop - reported by radiologist
Pain assessed by NRS 2 weeks after baseline | 2 weeks after baseline
  Patient pain level during the experience - reported by patient in a 10-level NRS

SECONDARY OUTCOMES:
Number of patients with bleeding despite 10 minutes compression | Baseline
  Bleeding despite 10 minutes compression - reported by radiologist
Radicality assessment fractions | Baseline
  Number of fractions possible to perform after the lesion has visually been removed - reported by radiologist
Self-reported number of patients who would recommend the procedure to others | 1 week after baseline
  Would the patient recommend the same procedure to others in same situation - reported by patient as yes or no
Self-reported satisfaction with cosmetic result assessed by a categorical scale | 1 week after baseline
  How dissatisfied is the patient with the cosmetic result - reported by patient - using a categorical scale from "not at all", "somewhat", "rather", "very".
Number of patients with self-reported occurrence of wound infection | 1 week after baseline
  Occurrence of wound infection - reported by patient as yes or no
Remaining scar | 6 months after baseline
  Yes = Any sign of prior trauma to the skin, No = Otherwise, Reported by radiologist as assessed by visual inspection
Pain assessed by NRS at baseline | At baseline
  Patient pain level during procedure - reported by patient in a 10-level NRS

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Strand, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No